CLINICAL TRIAL: NCT05493878
Title: Diagnostic Value of Tumor-Educated Platelets Integrin Alpha 2b (ITGA2B) and Selectin P (SELP) mRNA Expression in Pancreatic and Biliary Tract Cancer
Brief Title: ITGA2b and SELP Expression in Cancer Pancreas and Biliary Tract Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Hamdy Radwan, Doctor, Assiut University
Other Study IDs: TEPs genes in cancer pancrease
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Pancreas Cancer
Keywords: ITGA2b; SELP; Tumor educated platelets
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mRNA expression — Tumor educated platelets ITGA2b and SELP mRNA by reverse transcription-quantitative polymerase chain reaction (RT-qPCR).
  Other Names: gene expression; ITGA2b, SELP

SUMMARY:
1. To study the expression pattern of Integrin alpha 2b (ITGA2b) and Selectin P (SELP) genes of Tumor educated platelets in pancreatic and biliary tree cancer and its diagnostic value.
2. To investigate correlation between expression levels of ITGA2b and SELP genes and stages of pancreatic and biliary tree cancer.
3. To investigate correlation between expression levels of ITGA2b, SELP genes, CA 19-9 and CEA in pancreatic and biliary tree cancer patients.

DETAILED DESCRIPTION:
Malignant tumors arising in the biliary tract and pancreas are aggressive malignancies characterized by a poor prognosis and most of cases are diagnosed at advanced stages and have poor outcome . The most common pancreatic cancer is ductal adenocarcinoma, which accounts for about 80% of all pancreatic cancers. Pancreatic cancer is a highly lethal gastrointestinal cancer with a low 5-year survival rate and difficulty in early detection . Biliary tract cancers can be divided into intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer. CEA and CA 19-9 are the most common used serum biomarker for cancer screening and the diagnosis of pancreatic and biliary cancer.

Platelets are an essential component of the tumor microenvironment and serve as local and systemic respondents during tumor initiation and tumor metastasis. After interaction with tumor cells or tumor associated biomolecules, platelets can alter their RNA profile, and this process give rise to the so-called tumor educated platelets (TEPs). Tumor cells can directly and indirectly produce changes on platelet RNA and protein content, emerging a new term called liquid biopsy which reflect the presence of cancer and thus give hope to many that they might precede protein markers as a cancer-specific biomarker. Alterations in the TEPs RNA profile have been described as a novel source of potential biomarkers and can be used for early detection of cancer and treatment monitoring. Platelet biomarker transcripts can be transferred from tumor cells to platelets, although in some studies, the putative origin of the biomarker is the megakaryocyte (endogenous).

Integrin Alpha 2b (ITGA2b) gene encodes a member of the integrin alfa chain family of proteins which is proteolytically processed to form subunit of the alpha-IIb/beta-3 integrin cell adhesion receptor which is play crucial role in the blood coagulation system, by mediating platelets aggregation . Selectin P (SELP) gene encodes a protein that is stored in the alpha granules of platelets and Weibel-Palade bodies of endothelial cells. This protein redistributes to the plasma membrane during platelet activation and degranulation and mediates the interaction of activated endothelial cells or platelets with leukocytes. ITGA2b and SELP are cancer related genes and of the mRNA TEPs putative endogenous biomarkers which have a high value for detection of cancer, so, tumor educated platelets (TEPs) broadened the spectrum of liquid biopsy applications, and may enable blood-based cancer diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed pathologically as pancreatic and biliary cancer by gold standard test (pancreatic and biliary tract biopsy by endoscopy), male or female at any age.

Exclusion Criteria:

* History of anti-neoplastic therapy, such as chemotherapy or radiotherapy.
* Any other types of cancers.
* Any other clinically systemic acute or chronic inflammatory disease/s within one months.
* Autoimmune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at clinical pathology department, Assiut University Hospital, Faculty of medicine, Assiut University. Patient will be recruited from out patient clinics and in patients of the oncology department in Assiut university. Patients diagnosed pathologically as pancreatic and biliary cancer by gold standard test (pancreatic and biliary tract biopsy by endoscopy), male or female at any age
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Expression levels of ITGA2b and SELP on Tumor Educated PLatelets for diagnosis of pancreatic and biliary cancer | Baseline
  To study the expression pattern of ITGA2b and SELP genes of Tumor educated platelets in pancreatic and biliary tree cancer and its diagnostic value.

SECONDARY OUTCOMES:
Correlation between expression levels of ITGA2b and SELP on TEPs and the commonly used tumour marker CEA and CA 19-9 in the diagnosis of pancreatic and biliary cancer. | Baseline
  3- To investigate correlation between expression levels of ITGA2b, SELP genes, CA 19-9 and CEA in pancreatic and biliary tree cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ola A Afifi, doctor, Study Director — Ola A Afifi; Fatma M Helbawi, doctor, Study Chair — Fatma M Helbawi

REFERENCES:
- [Background] Xing S, Zeng T, Xue N, He Y, Lai YZ, Li HL, Huang Q, Chen SL, Liu WL. Development and Validation of Tumor-educated Blood Platelets Integrin Alpha 2b (ITGA2B) RNA for Diagnosis and Prognosis of Non-small-cell Lung Cancer through RNA-seq. Int J Biol Sci. 2019 Jul 24;15(9):1977-1992. doi: 10.7150/ijbs.36284. eCollection 2019. PMID 31523198
- [Background] D'Ambrosi S, Nilsson RJ, Wurdinger T. Platelets and tumor-associated RNA transfer. Blood. 2021 Jun 10;137(23):3181-3191. doi: 10.1182/blood.2019003978. PMID 33940602
- [Background] D'Ambrosi S, Visser A, Antunes-Ferreira M, Poutsma A, Giannoukakos S, Sol N, Sabrkhany S, Bahce I, Kuijpers MJE, Oude Egbrink MGA, Griffioen AW, Best MG, Koppers-Lalic D, Oudejans C, Wurdinger T. The Analysis of Platelet-Derived circRNA Repertoire as Potential Diagnostic Biomarker for Non-Small Cell Lung Cancer. Cancers (Basel). 2021 Sep 16;13(18):4644. doi: 10.3390/cancers13184644. PMID 34572871